CLINICAL TRIAL: NCT04194138
Title: Multi-Center Prospective Evaluation of Complex Adult Spinal Deformity Surgery
Brief Title: Complex Adult Deformity Surgery (CADS)
Acronym: CADS
Status: Recruiting | Type: Observational
Sponsor: International Spine Study Group Foundation (Other)
Collaborators: Medtronic (Industry); Globus Medical Inc (Industry); SI-BONE, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2123
Record Dates: First submitted 2019-11-25; First posted 2019-12-11 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Adult Spinal Deformity; Scoliosis; Kyphosis; Sagittal Imbalance
Keywords: Scoliosis; Kyphosis; Sagittal Imbalance; Spinal deformity
MeSH Terms: conditions — Scoliosis; Kyphosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Operative: A. Multicenter, prospective, nonrandomized analysis of operatively treated complex ASD patients meeting the following Inclusion Criteria
  1. 18 years of age or greater at the time of treatment
  2. Diagnosis of adult congenital, degenerative, idiopathic or iatrogenic spinal deformity
  3. Full body EOS radiographic assessment (sagittal and coronal visualization from skull to foot)
  4. Complex patients are defined as and meeting any one of the subsequent criteria:
     a. Radiographic criteria: i. PI-LL ≥ 25 degrees ii. TPA ≥ 30 degrees iii. SVA>15cm iv. Thoracic scoliosis ≥ 70 degrees v. Thoracolumbar/lumbar scoliosis ≥ 50 degrees vi. Global coronal malalignment >7cm b. Procedural criteria: i. Posterior spinal fusion > 12 levels ii. 3 column osteotomy or ACR c. Geriatric criteria: i. Age >65 years and minimum 7 levels of spinal instrumentation during surgery
  Interventions: Procedure: Index or spine revision surgery for complex adult spinal deformity

INTERVENTIONS:
Procedure: Index or spine revision surgery for complex adult spinal deformity — Surgical interventions will be patient specified by treating surgeon.

SUMMARY:
Evaluate surgical treatment outcomes and identify best practice guidelines for complex adult spinal deformity (ASD) patients, including radiographic and clinical outcomes, surgical and postoperative complications, risk factors for and revision surgery rates, and the role of standard work to improve patient outcomes and reduce surgical and postoperative complications.

DETAILED DESCRIPTION:
Specific Aims:

• Evaluate surgical treatment outcomes and identify best practice guidelines for complex adult spinal deformity (ASD) patients, including radiographic and clinical outcomes, surgical and postoperative complications, risk factors for and revision surgery rates, and the role of standard work to improve patient outcomes and reduce surgical and postoperative complications.

a. Complex ASD patients will be defined based upon clinical, radiographic and/or procedural criteria identified in an analysis of the existing ISSG ASD database: i. Magnitude of coronal and/or sagittal spinal deformity ≥75th percentile of patients in the ISSG database.

ii. Clinical or Radiographic parameters that corresponded to patients in the ISSG database that had complications requiring revision spine surgery and/or patients that had hospital length of stay >9 days.

iii. Procedures involving 3 column osteotomies and/or anterior column reconstruction (ACR) of the spine

* Develop and validate a standardized, universal complications classification system for spine surgery
* Evaluate perioperative blood management approaches, transfusion requirements, including variance in thresholds for blood transfusion and associated complications for adult spinal deformity surgery
* Assess impact of opioid use and pain management on patient cost, complications and outcomes
* Evaluate optimal opioid and analgesic usage and protocols for standard work development
* Evaluate clinical outcomes utilizing legacy patient reported outcome measures (PROMs) including modified Oswestry Disability Index (mODI), Scoliosis Research Society Questionnaire 22r (SRS-22r), Veterans RAND-12 (VR-12), and numeric pain rating scale (NRS) and compare the results of these legacy PROMs to outcomes scores as measured by the NIH Patient Reported Outcomes Measurement Information System (PROMIS) - PROMIS Anxiety, Depression, Pain Interference, Physical Function, and Social Satisfaction. Secondary aims for PROM research for this study include

  1. Validation of the PROMIS tool for ASD
  2. Establish a core set of PROMs for best practice guidelines for ASD
  3. Evaluate patient reported outcome variance for ASD according to SRS-Schwab spine deformity type including variance in baseline PROM domains impacted and variance in improvement in PROM domains
  4. Evaluate ASD outcomes compared to population norms and investigate/develop appropriate measures of clinically significant improvement
* Evaluate clinical outcomes stratifying by patient chronological and physiological age
* Evaluate measures to quantify patient physiological age including patient frailty for ASD and validate a frailty measurement system for ASD
* Evaluate the role of functional tests in patient's baseline frailty assessment including hand manometer and Edmonton Frail Scale. See appendix, pages 17 & 18 for details.
* Evaluate the contribution of patient frailty to patient outcomes, cost of care, disability, and complications
* Evaluate if patient frailty is a static measure or if frailty is a dynamic measure that can be improved through "pre-habilitation" and if the according associations with reductions in frailty correlate with reductions of cost, complications, and improvement in outcomes
* Evaluate cost variance for ASD surgery according to patient, institution, and geographical region and evaluate the cost effectiveness of surgical intervention for ASD
* Evaluate incidence of and risk factors for mental health (MH) compromise among ASD patients and establish best practice guidelines for assessing MH for ASD patients
* Evaluate the association of MH with surgical complications, outcomes, hospital length of stay and cost for ASD surgery
* Evaluate the association of social health surgical complications, outcomes, hospital length of stay and cost for ASD surgery and risk factors for routine (home) discharge vs. skilled nursing facility (SNF)/rehabilitation facility
* Broaden the evaluation of the surgically treated ASD patient to maximize evaluation of the entirety of the episode of care to include steps that can be taken prior to surgery including "prehabilitation," pain management, and MH care to improve treatment outcomes, reduce cost, reduce hospital length of stay, reduce non-routing discharge and reduce early and late complications
* Establish a core set of standard work guidelines to clinically and radiographically evaluate and treat ASD patients and evaluate the utility of standard work to improve outcomes for ASD and formulate best practice guidelines for surgical treatment of ASD
* Develop predictive analytic algorithms to risk stratify for best/worst outcomes, complications, sentinel events, and economic loss for ASD surgery

ELIGIBILITY:
Criteria:

Inclusion Criteria:

1. Diagnosis of adult congenital, degenerative, idiopathic or iatrogenic spinal deformity
2. Full body EOS radiographic assessment (sagittal and coronal visualization from skull to foot)
3. Complex patients are defined as and meeting any one of the subsequent criteria:

   1. Radiographic criteria:

      * PI-LL ≥ 25 degrees
      * TPA ≥ 30 degrees
      * SVA>15cm
      * Thoracic scoliosis ≥ 70 degrees
      * Thoracolumbar/lumbar scoliosis ≥ 50 degrees
      * Global coronal malalignment >7cm
   2. Procedural criteria:

      * Posterior spinal fusion > 12 levels
      * 3 column osteotomy or ACR
   3. Geriatric criteria:

      * Age >65 years and minimum 7 levels of spinal instrumentation during surgery

Exclusion Criteria:

1. Age <18 years of age
2. Active spine tumor or infection
3. Deformity due to acute trauma
4. Neuromuscular conditions/diseases (Parkinson's, Multiple Sclerosis, Post-polio syndrome)
5. Syndromic scoliosis
6. Inflammatory arthritis/auto immune diseases (Rheumatoid arthritis, Lupus, Ankylosing Spondylitis)
7. Prisoners
8. Women who are pregnant
9. Non English speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multi-center, prospective, non-randomized analysis of surgically treated complex adult spinal deformity (ASD) patients.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-07-30 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2032-07-31 (Estimated)

PRIMARY OUTCOMES:
Scoliosis Research Society (SRS) 22r | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Scoliosis specific patient reported outcome
Oswestry Disability Index (ODI) | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Spine specific patient reported outcome
Veterans RAND 12 Item Health Survey (VR-12) | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Patient reported outcome
Radiographic Evaluation | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Cobb angles, Coronal & Sagittal balance, spinopelvic measures
Patient-Reported Outcome Measurement Information System (PROMIS) - Anxiety | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Computer adaptive PROs
Patient-Reported Outcome Measurement Information System (PROMIS) - Depression | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Computer adaptive PRO
Patient-Reported Outcome Measurement Information System (PROMIS) - Pain Interference | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Computer adaptive PRO
Patient-Reported Outcome Measurement Information System (PROMIS) - Physical Function | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Computer adaptive PRO
Patient-Reported Outcome Measurement Information System (PROMIS) - Social Role Satisfaction | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Computer adaptive PRO
Patient-Reported Outcome Measurement Information System (PROMIS) - Social Satisfaction (DSA) | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Computer adaptive PRO
Visual Analog Scale - Back Pain | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Self-reported back pain on scale of 0 (No pain) to 10 (severe pain)
Visual Analog Scale - Leg Pain | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Self-reported leg pain on scale of 0 (No pain) to 10 (severe pain)

SECONDARY OUTCOMES:
Edmonton Frail Scale | Change from Preop to 3months and 1, 2, 5 & 10 year follow-up
  Evaluate frailty on scale of 0 to 17 where higher scores mean more frail
Canadian Study of Health and Aging (CSHA) | Change from Preop to 3months and 1, 2, 5 & 10 year follow-up
  Frailty scale of 1 to 8; higher scores mean more frail
Adverse Events | 3 months and 1, 2, 5 & 10 year post treatment
  Occurrence of Adverse events meeting reporting criteria and their relationship to intervention throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Shay Bess, MD, Principal Investigator — Denver International Spine Center; Lawrence Lenke, MD, Principal Investigator — Columbia University, Department of Orthopedic Surgery; Christopher Shaffrey, MD, Principal Investigator — Duke University, Departments of Neurosurgery and Orthopaedic Surgery
Locations (19):
- United States (18):
  - Shiley Center for Orthopaedic Research and Education at Scripps Clinic, La Jolla, California
  - University of California, Davis, Department of Orthopedic Surgery, Sacramento, California
  - UCSF, Department of Neurosurgery, San Francisco, California
  - Denver International Spine Center, Rocky Mountain Hospital for Children and Presbyterian St. Luke's Medical Center, Denver, Colorado
  - University of Kansas, Department of Orthopedic Surgery, Kansas City, Kansas
  - Norton Leatherman Spine Center, Louisville, Kentucky
  - Spine Institute of Louisiana, Shreveport, Louisiana
  - John Hopkins University, Department of Orthopedic Surgery, Baltimore, Maryland
  - Washington University, Department of Orthopedic Surgery, St Louis, Missouri
  - NYU, Department of Orthopedics, New York, New York
  - Hospital for Special Surgery, Department of Orthopedic Surgery, New York, New York
  - Columbia University Medical Center, New York, New York
  - Northwell Health, New York, New York
  - Duke University Health System, Durham, North Carolina
  - University Orthopedics, Providence, Rhode Island
  - Medical City Spine Hospital - Southwest Scoliosis Institute, Dallas, Texas
  - University of Texas - Houston, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
- Toronto Western, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Passias PG, Tretiakov P, Onafowokan OO, Das A, Lafage R, Smith JS, Line BG, Nayak P, Diebo B, Daniels AH, Gum JL, Hamilton DK, Buell TJ, Soroceanu A, Scheer JK, Eastlack RK, Mullin JP, Schoenfeld AJ, Mundis GM, Hosogane N, Yagi M, Mummaneni PV, Chou D, Fu KM, Than KD, Anand N, Okonkwo DO, Wang MY, Klineberg E, Kebaish KM, Lewis S, Hostin R, Gupta M, Lenke L, Kim HJ, Ames CP, Shaffrey CI, Bess S, Schwab F, Lafage V, Burton D. When is staging complex adult spinal deformity advantageous? Identifying subsets of patients who benefit from staged interventions. J Neurosurg Spine. 2024 Nov 22;42(2):185-192. doi: 10.3171/2024.8.SPINE24365. Print 2025 Feb 1. PMID 39576989